CLINICAL TRIAL: NCT03677674
Title: The Effects of Dehydration on the Performance of Judoka
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Laurent Chapelle, PhD student, Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: VrijeUniversiteitB
Record Dates: First submitted 2018-07-24; First posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Dehydration
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dehydrated (Experimental): The participants will be dehydrated (at least 2% of their body weight) before performing the Sterkowicz test.
  Interventions: Other: Dehydration
- euhydrated (No Intervention): The participants will be normally hydrated (= euhydration) before performing the Sterkowicz test (i.e. no specific intervention will be implemented).

INTERVENTIONS:
Other: Dehydration — Participants will be dehydrated (2% of their body weight) using sauna.
  Arms: dehydrated

SUMMARY:
Dehydration is a common phenomenon in judo that can lead to negative performance such as a decline in strength, a decline in anaerobic performance, a reduced body fluid balance, glycogen depletion and worsened psychological parameters. Therefore, we want to simulate several judo combats and look at the performances whether they change during a competition day. We also want to see if the results are different in a dehydrated versus euhydrated state.

ELIGIBILITY:
Inclusion Criteria:

* judoka
* minimum 18 years
* men and women
* only dehydration: sauna, warm bath, sweat suit

Exclusion Criteria:

* injured
* sick
* not underaged (18 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-12-20 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
Sterkowicz test | Up to 3 weeks
  Sterkowicz test

SECONDARY OUTCOMES:
heart rate | Up to 3 weeks
  Heart rate will be determined using the Polar H1 (Polar, Kempele, Finland)
Body weight | Up to 3 weeks
  Body weight will be assessed to the nearest 0.002 kg using the WLT 60/120/X/L3 scale (All Scales Europe, Veen, The Netherlands)
Borg Rating of Perceived Exertion Scale | Up to 3 weeks
  The Borg Rating of Perceived Exertion scale is a numerical scale (to determine exertion) that ranges from 6 to 20, where 6 means "no exertion at all" and 20 means "maximal exertion.
body temperature | Up to 3 weeks
  Body temperature will be determined using the Adtemp 421 Digital Ear Thermometer (American Diagnostics Corporations, Hauppauge, New York, United States of America)